CLINICAL TRIAL: NCT01616849
Title: Open-Label, Uncontrolled, Multicenter Phase II Study of Cisplatin and 5-Fu Combined With Nimotuzumab As First-Line Treatment in Patients With Untreated Metastatic Nasopharyngeal Carcinoma
Brief Title: Study of Chemotherapy Combined With Nimotuzumab in Untreated Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fujian Cancer Hospital (Other Government); First People's Hospital of Foshan (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Guangxi Medical University (Other); Guangzhou Medical University (Other); Hubei Cancer Hospital (Other); Hunan Provincial Cancer Hospital (Unknown); Hangzhou Cancer Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); Jiangxi Provincial Cancer Hospital (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); Wuhan University (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhao Chong, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PF-N-UMNPC
Record Dates: First submitted 2012-05-20; First posted 2012-06-12 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Stage IV Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PF+ Nimotuzumab (Experimental): Patients treated with cisplatin and 5-Fu combined with nimotuzumab
  Interventions: Drug: cisplatin and 5-Fu combined with nimotuzumab

INTERVENTIONS:
Drug: cisplatin and 5-Fu combined with nimotuzumab — DDP+5-Fu DDP 100 mg/m2 intravenous infusion in day1, 5-Fu 1000mg/m2/d continuous intravenous infusion on days 1 through 4, both drugs are given every 3 weeks.
  Nimotuzumab 200mg/d, intravenous infusion every week

SUMMARY:
This is an open-label, uncontrolled, multicenter phase II clinical trial. The purpose of this study is to evaluate acute toxicity and efficacy of cisplatin and 5-Fu combined with nimotuzumab in patients with untreated metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of nasopharyngeal carcinoma
* Distance metastasis at least 6 months after radical treatment
* Not suitable for local treatment, e.g. surgery, TACE
* At least one measurable lesion
* Estimate survival >3months
* Range from 18～70 years old
* PS 0~1
* WBC count ≥ 4×109/L，Hemoglobin ≥ 100g/L， platelet count ≥ 100×109/L
* ALT or AST < 2.5×ULN、bilirubin < 1.5×ULN
* 0Serum creatinine < 1.5×ULN

Exclusion Criteria:

* Central nervous system metastases
* Suitable for local treatment
* Second malignancy within 5 years
* Precious therapy with an investigational agent
* Uncontrolled seizure disorder or other serious neurologic disease
* ≥ Grade Ш allergic reaction to any drug including in this study
* Clinically significant cardiac or respiratory disease
* Creatinine clearance < 30ml/min
* Drug or alcohol addition
* Do not have full capacity for civil acts
* Severe complication, active infection
* Concurrent immunotherapy or hormone therapy for other diseases
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Objective response rate | study period of 19 Months
  To be determined by measurement of target lesions according to RECIST criteria
Progression free survival | 19 Months
  Defined as the time in months from first dose of Nimotuzumab until PD is observed or death occurs due to any cause.

SECONDARY OUTCOMES:
Overall survival | 19 Months
  Defined as the time in months from first dose of Nimotuzumab to the date of death is observed or to last follow-up visit.
Quality of life | 8 Months
  Using EORTC QLQ-C30(version 3.0) and EORTC QLQ-H&N35(Version 1.0) to access the quality of life. Collecting data before treatment, 1 week after each 2 cycles of chemotherapy, 1 months after all treatment finished.

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhao C, Miao J, Shen G, Li J, Shi M, Zhang N, Hu G, Chen X, Hu X, Wu S, Chen J, Shao X, Wang L, Han F, Mai H, Chua MLK, Xie C. Anti-epidermal growth factor receptor (EGFR) monoclonal antibody combined with cisplatin and 5-fluorouracil in patients with metastatic nasopharyngeal carcinoma after radical radiotherapy: a multicentre, open-label, phase II clinical trial. Ann Oncol. 2019 Apr 1;30(4):637-643. doi: 10.1093/annonc/mdz020. PMID 30689735
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn